CLINICAL TRIAL: NCT05538312
Title: AN INTERVENTIONAL, PHASE 1, OPEN-LABEL, FIXED SEQUENCE, 2-PERIOD STUDY TO ESTIMATE THE EFFECT OF MULTIPLE DOSES OF ITRACONAZOLE ON THE PHARMACOKINETICS OF SINGLE DOSE ARV-471 IN THE FED CONDITION IN HEALTHY ADULT MALES, AND FEMALES OF NONCHILDBEARING POTENTIAL
Brief Title: A Study to Understand the Effect of Itraconazole on the Levels of a Study Medicine Called ARV-471 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C4891009; 2022-003282-38 (EudraCT Number)
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vepdegestrant with and without itraconazole (Experimental): vepdegestrant administered as a single dose in Period 1 and Period 2. Itraconazole administered once a day for 11 days in Period 2.
  Interventions: Drug: vepdegestrant; Drug: Itraconazole

INTERVENTIONS:
Drug: vepdegestrant — Participants will receive a single dose of vepdegestrant by mouth in Period 1 and Period 2, with a washout period of at least 10 days between doses of vepdegestrant
  Other Names: ARV-471; PF-07850327
Drug: Itraconazole — Participants will receive itraconazole by mouth once a day for 11 days in Period 2.
  Other Names: Sporanox

SUMMARY:
The purpose of this study is to understand if a strong CYP3A4 inhibitor (itraconazole) affects how ARV-471 is processed and eliminated in healthy adults.

All participants in this study will receive one dose of ARV-471 alone by mouth in Period 1. In Period 2, everyone will receive itraconazole by mouth once a day for multiple days. Participants will also receive one dose of ARV-471 by mouth. The levels of ARV-471 in Period 1 will be compared to the levels of ARV-471 in Period 2 to determine if the CYP3A4 inhibitor affects how ARV-471 is processed differently in healthy adults.

ELIGIBILITY:
Inclusion Criteria

* Healthy male and/or female participants of non-childbearing potential who are overtly healthy as determined by medical evaluation including medical history, physical exam, laboratory tests, vital signs and standard 12-lead ECGs and are between the ages of 18 and 65 years, inclusive at the time of signing the informed consent document.
* Body Mass Index of 17.5 to 30.5 kg/meters squared; and a body weight >50 kg.
* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Pregnant female participants, breastfeeding female participants, female participants of childbearing potential.
* Male participants with partners currently pregnant; male participants who are unwilling or unable to use a highly effective method of contraception.
* Use of prescription or non-prescription medications, including vitamins, herbal and dietary supplements, grapefruit/grapefruit containing products, and Seville orange/Seville orange containing products within 7 days prior to the first dose of study intervention with the exception of:

Moderate/potent CYP3A inducers which are prohibited within 14 days plus 5 half-lives (whichever is longer) prior to the first dose of study intervention.

Moderate/potent CYP3A inhibitors which are prohibited within 14 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.

* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
* A positive urine drug test or alcohol breath test at discretion of investigator.
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest.
* Standard 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
* Aspartate transaminase or alanine aminotransferase level ≥ 1.0 × upper limit of normal.
* Total bilirubin level >1.0 × upper limit of normal; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ upper limit of normal.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
* History of use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes/day or 2 chews of tobacco/day.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* Known hypersensitivity or previous adverse events associated with azole antifungals or any of the formulation components of ARV-471.
* History of sensitivity to heparin or heparin induced thrombocytopenia.
* Estimated glomerular filtration rate <60 mL/min/1.73m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891009

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 periods in a single fixed sequence. A total of 12 participants were screened and enrolled into the study. All enrolled participants were treated and completed the study.
Groups:
- All Participants: Participants received a single dose of ARV-471 (PF-07850327) 200 milligram (mg) on Period 1 Day 1. After completion of Period 1, participants received 200 mg itraconazole once daily on Period 2 Days 1-4 and 6-11. On Period 2 Day 5, participants received a single dose of Itraconazole 200 mg first, immediately followed by a single dose of ARV-471 200 mg. Following Period 1, a washout period of at least 10 days must occur between the 2 single doses of ARV-471.
Period: Period 1 (6 Days)
Arm/Group | All Participants
Started | 12
Completed | 12
Not Completed | 0
Period: Period 2 (12 Days)
Arm/Group | All Participants
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline participants included all participants enrolled and who took at least 1 dose of study intervention.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.33 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUCinf) of ARV-471
Description: AUCinf was defined as area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUCinf) of ARV-471. AUCinf was calculated by AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: Period 1 Day 1: pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours post-dose; Period 2 Day 5: pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours post-dose
Population: Analysis population included all participants who received at least 1 dose of ARV-471 and/or itraconazole and had at least 1 of the ARV-471 or ARV-473 pharmacokinetic (PK) parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Period 1: ARV-471 200 mg: Participants received a single dose of ARV-471 200 mg on Period 1 Day 1.
- Period 2: ARV-471 200 mg + Itraconazole 200 mg: Participants received a single dose of Itraconazole 200 mg first, immediately followed by a single dose of ARV-471 200 mg on Period 2 Day 5.
Arm/Group | Period 1: ARV-471 200 mg | Period 2: ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
nanogram*hour per milliliter (ng*hr/mL) | 18960 (23) | 32020 (24)
Statistical Analysis 1: Comparison: Period 1: ARV-471 200 mg vs Period 2: ARV-471 200 mg + Itraconazole 200 mg; ARV-471 administered alone as Reference, ARV-471 administered after multiple doses of itraconazole as Test. Natural log transformed AUCinf was analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Other — Mixed Model; Ratio (%) of Adjusted Geometric Means = 168.90, 90% CI 2-sided [157.66 to 180.94] — The ratios (and 90% CIs) are expressed as percentages

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of ARV-471
Description: Cmax was defined as maximum plasma concentration. Cmax of ARV-471 was observed directly from data.
Time Frame: as for outcome 1
Population: Analysis population included all participants who received at least 1 dose of ARV-471 and/or itraconazole and had at least 1 of the ARV-471 or ARV-473 PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Period 1: ARV-471 200 mg | Period 2: ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
nanogram per milliliter (ng/mL) | 517.9 (22) | 788.2 (19)
Statistical Analysis 1: Comparison: Period 1: ARV-471 200 mg vs Period 2: ARV-471 200 mg + Itraconazole 200 mg; ARV-471 administered alone as Reference, ARV-471 administered after multiple doses of itraconazole as Test. Natural log transformed Cmax was analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Other — Mixed Model; Ratio (%) of Adjusted Geometric Means = 152.19, 90% CI 2-sided [136.90 to 169.18] — The ratios (and 90% CIs) are expressed as percentages

3. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to 120 Hours (AUC120) of ARV-473
Description: ARV-473 was the epimer of ARV-471. AUC120 was defined as area under the plasma concentrationtime profile from time zero to 120 hours. AUC120 was calculate by Linear/Log trapezoidal method.
Time Frame: Period 1 Day 1: pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours post-dose; Period 2 Day 5: pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 1: ARV-471 200 mg | Period 2: ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 4734 (30) | 7668 (28)
Statistical Analysis 1: Comparison: Period 1: ARV-471 200 mg vs Period 2: ARV-471 200 mg + Itraconazole 200 mg; ARV-471 administered alone as Reference, ARV-471 administered after multiple doses of itraconazole as Test. Natural log transformed AUC120 was analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Other — Mixed Model; Ratio (%) of Adjusted Geometric Means = 161.99, 90% CI 2-sided [148.70 to 176.47] — The ratios (and 90% CIs) are expressed as percentages

4. Primary Outcome: Cmax of ARV-473
Description: ARV-473 was the epimer of ARV-471. Cmax was defined as maximum plasma concentration. Cmax of ARV-473 was observed directly from data.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 1: ARV-471 200 mg | Period 2: ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
ng/mL | 56.37 (26) | 86.31 (27)
Statistical Analysis 1: Comparison: Period 1: ARV-471 200 mg vs Period 2: ARV-471 200 mg + Itraconazole 200 mg; [analysis description as in outcome 2, analysis 1]; Test type: Other — Mixed Model; Ratio (%) of Adjusted Geometric Means = 153.13, 90% CI 2-sided [138.51 to 169.30] — The ratios (and 90% CIs) are expressed as percentages

5. Secondary Outcome: Area Under the Plasma Concentration Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of ARV-471
Description: AUClast was defined as area under the plasma concentrationtime profile from time zero to the time of the last quantifiable concentration (Clast). AUClast was calculated by Linear/Log trapezoidal method.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 1: ARV-471 200 mg | Period 2: ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 16730 (24) | 28710 (21)
Statistical Analysis 1: Comparison: Period 1: ARV-471 200 mg vs Period 2: ARV-471 200 mg + Itraconazole 200 mg; ARV-471 administered alone as Reference, ARV-471 administered after multiple doses of itraconazole as Test. Natural log transformed AUClast was analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% CIs were obtained from the model and were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Other — Mixed Model; Ratio (%) of Adjusted Geometric Means = 171.63, 90% CI 2-sided [159.96 to 184.15] — The ratios (and 90% CIs) are expressed as percentages

6. Secondary Outcome: AUC120 of ARV-471
Description: AUC120 was defined as area under the plasma concentrationtime profile from time zero to 120 hours. AUC120 was calculate by Linear/Log trapezoidal method.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 1: ARV-471 200 mg | Period 2: ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 16730 (24) | 26400 (20)
Statistical Analysis 1: Comparison: Period 1: ARV-471 200 mg vs Period 2: ARV-471 200 mg + Itraconazole 200 mg; [analysis description as in outcome 3, analysis 1]; Test type: Other — Mixed Model; Ratio (%) of Adjusted Geometric Means = 157.80, 90% CI 2-sided [146.51 to 169.95] — The ratios (and 90% CIs) are expressed as percentages

7. Secondary Outcome: Time for Cmax (Tmax) of ARV-471
Description: Time for Cmax of ARV-471 was observed directly from data as time of first occurrence.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Period 1: ARV-471 200 mg | Period 2: ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
hour | 6.00 [2.00 to 8.00] | 6.00 [4.00 to 8.00]

8. Secondary Outcome: Terminal Half-Life (t1/2) of ARV-471
Description: Terminal half-life (t1/2) was calculated by Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Period 1: ARV-471 200 mg | Period 2: ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
hour | 42.64 (4.0800) | 61.57 (9.1196)

9. Secondary Outcome: Apparent Clearance After Oral Dose (CL/F) of ARV-471
Description: CL/F was defined as apparent oral clearance and calculated by dose/AUCinf. AUCinf was defined as area under the plasma concentration-time curve from time 0 extrapolated to infinite time.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | Period 1: ARV-471 200 mg | Period 2: ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
liter per hour (L/hr) | 10.54 (23) | 6.245 (24)

10. Secondary Outcome: Apparent Volume of Distribution After Oral Dose (Vz/F) of ARV-471
Description: Vz/F was defined as apparent volume of distribution calculated by dose/(AUCinf * kel). AUCinf was defined as area under the plasma concentration-time curve from time 0 extrapolated to infinite time and kel was defined as the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Period 1: ARV-471 200 mg | Period 2: ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
liter (L) | 645.6 (29) | 549.5 (20)

11. Secondary Outcome: AUClast of ARV-473
Description: ARV-473 was the epimer of ARV-471. AUClast was defined as area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (Clast). AUClast was calculated by Linear/Log trapezoidal method.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 1: ARV-471 200 mg | Period 2: ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 4734 (30) | 9129 (31)
Statistical Analysis 1: Comparison: Period 1: ARV-471 200 mg vs Period 2: ARV-471 200 mg + Itraconazole 200 mg; [analysis description as in outcome 5, analysis 1]; Test type: Other — Mixed Model; Ratio (%) of Adjusted Geometric Means = 192.86, 90% CI 2-sided [178.86 to 207.94] — The ratios (and 90% CIs) are expressed as percentages

12. Secondary Outcome: Tmax of ARV-473
Description: ARV-473 was the epimer of ARV-471. Time for Cmax of ARV-473 was observed directly from data as time of first occurrence.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Period 1: ARV-471 200 mg | Period 2: ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
hour | 24.0 [24.0 to 48.1] | 35.9 [12.0 to 47.8]

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship with the study intervention. SAE is defined as one of the following: is fatal or life threatening; results in persistent or significant disability/incapacity; constitutes a congenital anomaly/birth defect; is medically significant; requires inpatient hospitalization or prolongation of existing hospitalization. Treatment-emergent AE is defined as an AE with onset date occurring during the on-treatment period. AEs include all SAEs and non-SAEs.
Time Frame: From the first dose (Day 1) up to 35 days after the last dose of study intervention (up to 52 days)
Population: All participants enrolled and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- ARV-471 200 mg: Participants received a single dose of ARV-471 200 mg on Day 1 of Period 1.
- Itraconazole 200 mg: Participants received itraconazole 200 mg once daily alone over a period of Days 1-4 in Period 2.
- ARV-471 200 mg + Itraconazole 200 mg: Participants received a single dose of ARV-471 200 mg on Day 5 of Period 2 co-administered with itraconazole 200 mg once daily on Days 5-11 in Period 2.
Arm/Group | ARV-471 200 mg | Itraconazole 200 mg | ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12 | 12
Participants
  Treatment-emergent AEs | 2 | 3 | 2
  Treatment-emergent SAEs | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); liver function (aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine, uric acid, cystatinC); electrolytes (sodium, potassium, chloride, calcium, bicarbonate); clinical chemistry (glucose); urinalysis (dipstick [decimal logarithm of reciprocal of hydrogen ion activity {pH} of urine, glucose, protein, blood, ketones, nitrites, leukoesterase, urobilinogen, bilirubin], microscopy. Abnormality was determined at the investigator's discretion.
Time Frame: Baseline (Period 1 Day -1) up to Period 2 Day 12 (19 days)
Population: All participants enrolled and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | ARV-471 200 mg | ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
Participants | 4 | 1

15. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs (blood pressure and pulse rate) were obtained with participant following at least a 5-minute rest in a supine position. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: Baseline (Period 1 Day 1) up to Period 2 Day 5 (11 days)
Population: All participants enrolled and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | ARV-471 200 mg | ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: ECG abnormalities criteria include a) a postdose QTc corrected using Fridericia's formula (QTcF) increased by ≥60 millisecond (ms) from the baseline and the absolute QTcF value >450 ms; or b) an absolute QTcF value ≥500 ms for any scheduled ECG.
Time Frame: Baseline (Period 1 Day 1) up to Period 2 Day 12 (18 days)
Population: All participants enrolled and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | ARV-471 200 mg | ARV-471 200 mg + Itraconazole 200 mg
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose (Day 1) up to 35 days after the last dose of study intervention (up to 52 days).
Arm/Group | ARV-471 200 mg | Itraconazole 200 mg | ARV-471 200 mg + Itraconazole 200 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 3/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ARV-471 200 mg (N=12) | Itraconazole 200 mg (N=12) | ARV-471 200 mg + Itraconazole 200 mg (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Gingival discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
AUCinf for ARV-473 could only be reported for 2 of 12 participants in Period 1 (ARV-471 alone) and 6 of 12 participants in Period 2 (ARV-471 + itraconazole) based on protocol prespecified criteria, therefore was not used as the primary endpoint for ARV-473. Furthermore, AUC120, was selected as the primary endpoint for ARV-473 in lieu of AUClast to account for the difference in sampling intervals between Test Treatment (0-168 hours) and Reference Treatment (0-120 hours).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT05538312/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT05538312/SAP_001.pdf